CLINICAL TRIAL: NCT06819735
Title: A Phase 1/2, Multicentre, Open-label Clinical Trial of DT-7012 as Monotherapy and in Combination With an Immune Checkpoint Inhibitor in Participants With Selected Advanced Solid Tumors (DOMISOL, DOmain_therapeutics Monoclonal antIbody for SOLid Tumors)
Brief Title: Study of DT-7012 as a Single Agent and in Combination With an Immune Checkpoint Inhibitor in Participants With Advanced Solid Tumors
Acronym: DOMISOL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Domain Therapeutics Australia Pty Ltd (Industry)
Collaborators: Domain Therapeutics SA (Industry)
Responsible Party: Sponsor
Organization: Domain Therapeutics SA (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DT-7012-CLI-001
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1A (Experimental): Dose escalation of DT-7012 as a single agent
  Interventions: Drug: DT-7012
- Part 1B (Experimental): Dose escalation of DT-7012 in combination with an ICI
  Interventions: Drug: DT-7012; Drug: Immune checkpoint inhibitor
- Phase 2 (Experimental): Evaluation of DT-7012 as a sinle agent and/or in combination with an immune checkpoint inhibitor in indication-specific cohorts.
  Interventions: Drug: DT-7012; Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: DT-7012 — Intravenous infusion
Drug: Immune checkpoint inhibitor — Intravenous infusion
  Arms: Part 1B; Phase 2

SUMMARY:
This is a phase 1/2, dose-escalation, clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of DT-7012 (an anti-CCR8 monoclonal antibody) as a single agent and in combination with an immune checkpoint inhibitor in adult participants with selected advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase 1/2, first-in-human, multicenter, open-label clinical study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of DT-7012, administered as monotherapy and in combination with an immune checkpoint inhibitor (ICI), in participants with selected recurrent advanced/metastatic solid tumors.

This study includes:

* a phase 1 Monotherapy Dose Escalation
* a phase 1b Combination Dose Escalation (this part will be initiated upon recommendation from the Safety Review Committee based on Monotherapy Dose Escalation data and corresponds to a dose escalation of a combination of DT-7012 with an ICI)
* a subsequent phase 2 Indication-Specific Efficacy part

The phase 1 aims at determining the maximum tolerated dose or maximum administered dose of DT-7012 as single agent and in combination with an ICI, and the safety and tolerability of DT-7012 as single agent and in combination with an ICI in participants with selected recurrent advanced/metastatic solid tumors.

The phase 2 will assess the efficacy of DT-7012 as monotherapy and/or in combination with an ICI in indication-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor, among selected cancer types, that is recurrent, locally advanced (i.e., not eligible for curative surgery or radiotherapy) or metastatic, has progressed after at least one line of systemic therapy and has no established curative option.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed by the local site investigator/radiologist.
* At least 1 tumour lesion accessible to biopsy per treating physician judgement.
* Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
* Adequate organ function.

Exclusion Criteria:

* Any unresolved AEs from previous anti-cancer therapies of grade ≥2, with the exception of alopecia.
* Prior severe immune-related AEs (irAEs) leading to immunotherapy treatment discontinuation.
* Major surgery or significant traumatic injury within 4 weeks prior to Cycle 1 Day 1 with unadequately recovered AEs and/or complications from the intervention prior to Cycle 1 Day 1.
* Prior radiotherapy within the 4 weeks prior to Cycle 1 Day 1 or limited field palliative radiotherapy within 2 weeks prior to Cycle 1 Day 1.
* Prior anti-CCR8 monoclonal antibody treatment received in an investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with DLTs, TEAEs, TRAEs, AESIs, SAEs and AEs leading to treatment discontinuation | Cycle 1 (21 days)
  Proportion of participants with dose-limiting toxicities (DLTs), treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), adverse events of special interest (AESIs), serious adverse events (SAEs) and adverse events (AEs) leading to treatment discontinuation

SECONDARY OUTCOMES:
Objective response rate (ORR) | From the first dose of study drug until the date of disease progression/recurrence, assessed up to 12 months
  The anti-tumor activity will be determined based on the assessment of, but not limited to, the objective response rate (ORR). ORR is defined as the percentage of participants with a complete response (CR) or a partial response (PR) at any time during the study according to RECIST v1.1 and immune RECIST (iRECIST) as assessed by the investigator.
Serum concentrations of DT-7012 | From the first dose of study drug until the date of end of treatment, assessed up to 12 months
  Serum concentrations of DT-7012 will be determined to evaluate the pharmacokinetics (PK) of DT-7012

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Macquarie University Clinical Trial Unit, North Ryde, New South Wales
  - Cancer Research SA, Adelaide, South Australia
  - Peninsula & South Eastern Haematology & Oncology Group, Frankston, Victoria
  - Cabrini Health Limited, Malvern, Victoria
  - One Clinical Research Pty Ltd, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No